CLINICAL TRIAL: NCT04928001
Title: A Feasibility Study for Implementing and Evaluating an Internet-based Cognitive Behavior Therapy Intervention in School Settings and Its Impact on Adolescent Mental and Behavioral Health
Brief Title: Implementing and Evaluating an Internet-based Cognitive Behavior Therapy Intervention in School Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Principal Investigator, Kathryn Franklin, Assistant Teaching Professor, Montana State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KF072420
Record Dates: First submitted 2021-06-09; First posted 2021-06-16 (Actual); Results first posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: Depression Anxiety and Co-occurring Rural Youth

STUDY DESIGN:
Intervention Model Description: multiple baseline pre-post design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth Thrive iCBT program (Other): Youth Thrive iCBT online program
  Interventions: Other: internet based iCBT program, Youth Thrive

INTERVENTIONS:
Other: internet based iCBT program, Youth Thrive — iCBT program is a skills program which teaches assertive communication, constructive thinking and rewarding activities

SUMMARY:
This research study examines rural youth's experience of an internet based cognitive behavioral therapy intervention, and their experience of symptoms of depression, anxiety and co-occurring disorders.

DETAILED DESCRIPTION:
In the United States, and rural Montana, a substantial health disparity exists for rural youths' mental health and mental health care access. In 2017, nearly a third of all Montana high school students reported being impacted by depression; 21% considered suicide compared to 17% nationally. Over 30% of Montana adolescents indicated drinking alcohol and 20% indicated using marijuana. Rural Montanans face enormous barriers to behavioral health care including low mental health care provider coverage, long distances to adequate care, and stigma. We have developed a culturally and developmentally appropriate Internet-based Cognitive Behavior Therapy (iCBT) program designed to teach skills that address mental and behavioral health challenges common to adolescents. Building on previous development and evaluation of an adult version of iCBT (Thrive), the investigators propose to pilot the newly developed youth version of Thrive (Y-T), a fully automated stand-alone program. Y-T will deliver CBT skills through educational, real life adolescent scenarios, and tailored feedback videos to address symptoms of depression, anxiety and co-occurring (addiction) behaviors. The investigators intend to conduct feasibility analyses of pilot study implementation in school communities. The investigators will document and assess organization-level facilitators and barriers that impact the study processes at each study site. Short-term goal for this research are to understand how to effectively conduct trials within school community settings and to obtain preliminary information on the acceptability and effectiveness of the Y-T program to address depression and anxiety symptoms, and addictive behaviors. The investigators will conduct post-intervention focus groups to assess the program as experienced by participants and insight on the extent of program engagement and learning. The investigators hypothesize that those using Y-T over an 8-week period will report markedly decreased scores on anxiety, depression, and addictive behaviors. The long-term goal is to conduct a larger trial of the program to determine the evidence of impact among youth. Provided that this research demonstrates such programs to be evidence-based, the investigators will work on a broader dissemination plan with the ultimate aim of decreasing mental and behavioral health and respective health care disparities among rural youth.

ELIGIBILITY:
Inclusion Criteria:

* participants are youth enrolled in participating schools
* ages 13 - 18 years old
* have access to electronic device to access iCBT intervention

Exclusion Criteria:

* none.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montana State University, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Franklin K, Tribbit T. A Feasibility Study for Implementing and Evaluating an Internet-Based Cognitive Behavior Therapy Intervention in Rural School Settings and its Impact on Adolescent Mental and Behavioral Health. Chronicle of Rural Education. 2024; 2(1).
- See also: Link to published article and results — https://ojs.library.okstate.edu/osu/index.php/chronicle-of-rural-education/article/view/9566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Youth Thrive iCBT Program
Started | 67
Completed | 47
Not Completed | 20

BASELINE CHARACTERISTICS:
Population: Inclusion Criteria:
  participants are youth enrolled in participating schools ages 13 - 18 years old have access to electronic device to access iCBT intervention
Arm/Group | Youth Thrive iCBT Program
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  Depressive Symptoms: <=18 years | 67
  Depressive Symptoms: Between 18 and 65 years | 0
  Depressive Symptoms: >=65 years | 0
  Anxiety Symptoms: <=18 years | 67
  Anxiety Symptoms: Between 18 and 65 years | 0
  Anxiety Symptoms: >=65 years | 0
  Substance Use Attitudes & Behaviors: <=18 years | 67
  Substance Use Attitudes & Behaviors: Between 18 and 65 years | 0
  Substance Use Attitudes & Behaviors: >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Beck's Anxiety Inventory, Youth Version
Description: The inventory measures anxiety symptoms and utilizes T Scores. 52.45 indicates the population mean with a standard deviation of 11.4 55 or less minimal, average symptoms of anxiety 55-59 mild symptoms of anxiety 60-69 moderate symptoms of anxiety 70+ severe symptoms of anxiety
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Youth Thrive iCBT Program
Number analyzed (Participants) | 67
T Score | 52.45 (11.4)
Statistical Analysis 1: Comparison: Youth Thrive iCBT Program; Test type: Superiority; p = .01, t-test, 1 sided; Mean Difference (Final Values) = 31, 95% CI 2-sided [0 to 60]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Youth Thrive iCBT Program
All-Cause Mortality (participants affected / at risk) | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT04928001/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT04928001/ICF_001.pdf